CLINICAL TRIAL: NCT06935903
Title: Assessment of Physical Capacity and Metabolic Parameters in Marathon Runners With Type 1 Diabetes: an Observational Study
Brief Title: Marathon Runners With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zozulińska-Ziółkiewicz Dorota MD PhD, Head of the Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences
Other Study IDs: NdS/544750/2021/2022; 1245/18 (Other: Ethical Committee of Poznan University of Medical Sciences)
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 Diabetes; Physical Activity; Physical Endurance; Absorptiometry; Oxygen Consumption
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Type 1 diabetes group: Male participants with confirmed T1DM diagnosis for ≥1 year who have completed a marathon.
- Control Group: Healthy male marathon runners matched by age, sex, and training background

SUMMARY:
The goal of this observational study is to learn about the physical capacity and metabolic characteristics of male marathon runners with type 1 diabetes mellitus (T1DM). The main question it aims to answer is:

Do male marathon runners with T1DM have different physical fitness and metabolic profiles compared to healthy runners without diabetes?

Participants with T1DM and healthy controls who have completed a marathon will undergo a single in-person assessment, including body composition analysis, resting metabolic rate measurement, and a maximal exercise test

DETAILED DESCRIPTION:
This observational, cross-sectional case-control study aims to compare physical capacity and metabolic parameters between male marathon runners with type 1 diabetes mellitus (T1DM) and healthy male marathon runners without diabetes. The study focuses on evaluating differences in cardiopulmonary fitness, resting metabolic rate, and body composition between the two groups.

Participants attended a single study visit after overnight fasting. The visit included anthropometric measurements, assessment of medical history, and structured questionnaires on diabetes management (for T1DM participants) and physical activity habits. Body composition was assessed using dual-energy X-ray absorptiometry (DXA), providing detailed analysis of total and regional fat mass, lean tissue mass, and bone mineral density. Daily calibration of the DXA scanner ensured data accuracy and consistency.

Resting metabolic rate (RMR) was measured by indirect calorimetry using a ventilated hood system. Measurements were performed in a controlled environment with standardized temperature and low light to minimize variability. Data collection spanned 25 minutes, with the first 5 minutes discarded for acclimatization and the subsequent 20 minutes analyzed. Energy expenditure and substrate oxidation rates were calculated using established equations (Weir equation and Zuntz table).

Cardiorespiratory fitness was assessed through a maximal exercise test on a cycle ergometer with continuous respiratory gas analysis. The test protocol began with a resting phase and warm-up, followed by incremental workload increases until volitional exhaustion. Parameters such as VO₂max, ventilatory efficiency, gas exchange threshold, and peak workload were measured using a calibrated metabolic cart.

Data analysis involved descriptive statistics, Mann-Whitney U tests for numerical comparisons, and Chi-square tests for categorical variables. Dedicated manufacturer software was used for CPET data processing, and statistical analyses were conducted using R software (version 4.4.1).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of T1DM for at least 1 year.
* Age ≥ 18 years.
* Written informed consent and adherence to the study protocol.

Exclusion Criteria:

* Pregnancy.
* Use of medications significantly affecting metabolism or exercise performance
* Presence of chronic medical or psychiatric conditions limiting safe participation

  •Presence of advanced chronic complications of diabetes: proliferative retinopathy, diabetic kidney disease in stages III-V, cardiovascular diseases
* Inability to safely complete maximal exercise testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult marathon runners aged ≥18 years. Participants in the T1DM group with a confirmed diagnosis of T1DM for at least one year. The control group comprises healthy people with similar physical activity levels but no chronic health conditions.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
VO₂max (mL/kg/min) | single visit
  peak oxygen uptake during graded exercise testing

SECONDARY OUTCOMES:
Resting metabolic rate (kcal/day) | single visit
  The amount of energy expended by the body at rest in a fasting state, measured in kilocalories per day using indirect calorimetry.
Body adipose percentage [%] | single visit
  The proportion of a person's total body mass that is composed of adipose tissue, assessed using dual-energy X-ray absorptiometry (DXA).
Lean tissue percentage [%] | single visit
  The proportion of a person's total body mass that is composed of lean tissue, assessed using dual-energy X-ray absorptiometry (DXA).
Forced Vital Capacity [L] | single visit
  the total volume of air exhaled forcefully after a full inhalation, measured in liters.
Maximum Vital Capacity [L] | single visit
  the greatest volume of air that can be exhaled after a maximal inhalation, measured in liters.
Forced Expiratory Volume in 1 second [%] | single visit
  the percentage of the Forced Vital Capacity that is exhaled during the first second of a forced breath, indicating airway function

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Zozulinska-Ziolkiewicz, MD, PhD, Principal Investigator — Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences
Locations (1):
- Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the small sample size and the potential risk of participant re-identification, even with de-identified data. The study was not designed with broad data sharing in mind, and no participant consent was obtained for public data release.

REFERENCES:
- [Background] Shepherd JA, Ng BK, Sommer MJ, Heymsfield SB. Body composition by DXA. Bone. 2017 Nov;104:101-105. doi: 10.1016/j.bone.2017.06.010. Epub 2017 Jun 16. PMID 28625918
- [Background] Achamrah N, Delsoglio M, De Waele E, Berger MM, Pichard C. Indirect calorimetry: The 6 main issues. Clin Nutr. 2021 Jan;40(1):4-14. doi: 10.1016/j.clnu.2020.06.024. Epub 2020 Jul 2. PMID 32709554
- [Background] Poole DC, Wilkerson DP, Jones AM. Validity of criteria for establishing maximal O2 uptake during ramp exercise tests. Eur J Appl Physiol. 2008 Mar;102(4):403-10. doi: 10.1007/s00421-007-0596-3. Epub 2007 Oct 30. PMID 17968581
- [Background] Thuillier P, Domun N, Sonnet E, Le Ven F, Roudaut C, Kergus A, Kerlan V, Roudaut N. Prevention of exercise-induced hypoglycemia in 12 patients with type 1 diabetes running the Paris Marathon using continuous glucose monitoring: A prospective, single-center observational study. Diabetes Metab. 2022 Mar;48(2):101321. doi: 10.1016/j.diabet.2022.101321. Epub 2022 Jan 12. PMID 35032674
- [Background] Grimm JJ, Muchnick S. Type I diabetes and marathon running. Diabetes Care. 1993 Dec;16(12):1624. doi: 10.2337/diacare.16.12.1624a. No abstract available. PMID 8299461
- [Background] Riddell MC, Scott SN, Fournier PA, Colberg SR, Gallen IW, Moser O, Stettler C, Yardley JE, Zaharieva DP, Adolfsson P, Bracken RM. The competitive athlete with type 1 diabetes. Diabetologia. 2020 Aug;63(8):1475-1490. doi: 10.1007/s00125-020-05183-8. Epub 2020 Jun 12. PMID 32533229
- [Background] Chimen M, Kennedy A, Nirantharakumar K, Pang TT, Andrews R, Narendran P. What are the health benefits of physical activity in type 1 diabetes mellitus? A literature review. Diabetologia. 2012 Mar;55(3):542-51. doi: 10.1007/s00125-011-2403-2. Epub 2011 Dec 22. PMID 22189486
- See also: Poznan University of Medical Sciences in Poznań is conducting the project "Development of the University Centre for Sports and Medical Studies in Poznań" (No. NdS/544750/2021/2022), funded by the Ministry of Education and Science under th — https://ucbsm.ump.edu.pl/nauka-dla-spoleczenstwa